TITLE: The R-CITY Project: A Collaborative Intervention with Teachers and Youth

**NCT #: SBS2232** 

**VERSION DATE: September 10, 2021** 

**Study Title:** The R-CITY Project **Version Date:** V5, 8/19/2021

University of Virginia Principal Investigator: Catherine Bradshaw, Ph.D.

University of Virginia IRB No: #2232

# **Informed Consent Agreement**

### **R-CITY Coaching Consent Form for School Staff**

Please read this consent agreement carefully before you decide to participate in the study.

#### **Consent Form Key Information:**

- You are being asked to join a research study.
- University of Virginia is leading this study.
- This consent form explains the research study and your part in the study.
- Please read it carefully and take as much time as you need.
- Your participation is voluntary. You can choose not to participate. If you join, you may quit at any time with no penalty.
- During the study, you will be informed regarding any new information that might affect your decision to continue in the study.

**Purpose of the research study:** The project is designed to support and enhance the implementation of the Second Step social-emotional learning curriculum initiative in Anne Arundel County Public Schools. Coaches will provide supports to teachers implementing the social emotional learning curriculum in their classrooms. In addition, coaches will provide school wide professional development, 1:1 coaching for participating teachers, and an additional set of six student lessons designed to promote teacher and student skills in equity literacy and teachers' use of culturally responsive teaching practices. In this project, equity means providing all people the resources and treatment that gives them a fair chance to succeed. Equity literacy refers to the knowledge and skills to ensure and advocate for equity in ones' spheres of influence. The project's supports and enhancements are being tested through a *school* randomized controlled trial. This means that the principal at your school agreed to have the school participate and understands that the *whole school* will be randomly selected to receive ONE of two project conditions:

- 1) "Classroom", which includes school and teacher supports from project coaches to enhance implementation of the Second Step program, a teacher-led, classroom-based social emotional learning curriculum provided by Anne Arundel County Public Schools; OR
- 2) "Classroom *Plus*", which includes school and teacher supports from project coaches to enhance implementation of the Second Step program, plus additional professional

development and 1:1 coaching for teachers, and six teacher-led equity literacy lessons for students.

As a classroom teacher at a participating R-CITY school, you are being asked to participate in this research study.

**What you will do in the study:** R-CITY schools will be *randomly selected* to either the Classroom or Classroom *Plus* condition.

If your school is *randomly* selected to the *Classroom* condition, we will ask that you:

- Communicate with a project coach on SEL curriculum implementation supports as needed.
- Allow members of the research study to conduct non-evaluative classroom observations during instruction.
- Complete online self-report surveys at 2 time points (fall and spring of current school year) about your knowledge, skills, and self-efficacy related to implementing the Second Step lessons in your classroom. We will also ask for your demographic information, including teacher age, household income, gender, race/ethnicity, role in school, and number of years working in the school. This is to help us understand other factors that may influence the effects of this intervention.

If your school is *randomly* selected to the <u>Classroom Plus</u> condition, we will ask that you do the above *plus*:

- Participate in an initial Teacher Interview with a project coach.
- Allow additional classroom observations by the project coach and meet with the coach to discuss feedback.
- Implement six equity literacy lessons in your classroom, including receiving implementation support from coaches and participating in a 90-minute training in the curriculum.

**Time required:** The study will require at least 1 hour and 20 minutes hour of your time, including completing the self-report survey (20 minutes) and participating in supports for implementing your school's SEL curriculum (1 hour). If your school is randomized to the Classroom *Plus* condition, the study will require an additional 7.5 hours of your time. This includes approximately 3 hours for one-on-one coaching, 3 hours of equity literacy lesson implementation during regularly scheduled class time, and 1.5 hours of training.

**Risks:** There is a small possibility that you may feel pressured to provide certain kinds of responses on your self-report survey. Therefore, you will complete the survey confidentially online using a personal identification (or ID) code to safeguard the confidentiality of your responses with the survey materials.

**Benefits:** You will receive training, experience, and support in the delivery of the Second Step curriculum as well as in implementing equity literacy lessons and content to your students.

The study may help us identify factors that improve classroom equity, classroom management skills, student engagement, and reduce discipline disproportionality.

Confidentiality: This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you unless you say it is okay. Your information will be assigned a code number. The list connecting your name to this code will be kept in a locked file. When the study is completed and the data have been analyzed, this list will be destroyed. Your name will not be used in any report. You can have access to and release information about your research involvement.

Voluntary participation: Your participation in the study is completely voluntary.

**Right to withdraw from the study:** You have the right to withdraw from the study at any time without penalty.

How to withdraw from the study: There is no penalty for withdrawing. If you would like to withdraw from the study, please contact Dr. Catherine Bradshaw at cpb8g@virginia.edu.

Payment: You will receive a \$25 gift card for your completion of each self-report survey.

Using data beyond this study: This study was funded by the National Institute of Minority Health and Health Disparities (NIMHD) and de-identified data may be archived. Your identity will not be in files shared with the NIMHD.

### If you have questions about the study, contact:

Catherine P. Bradshaw, Ph.D., M.Ed. Professor and R-CITY Principal Investigator Curry School of Education & Human Development University of Virginia, PO Box 400260 Charlottesville, VA 22904

Telephone: (434) 924-8121

Email address: cpb8g@virginia.edu

To obtain more information about the study, ask questions about the research procedures, express concerns about your participation, or report illness, injury or other problems, please contact:

Tonya R. Moon, Ph.D.

Chair, Institutional Review Board for the Social and Behavioral Sciences

One Morton Dr Suite 500

University of Virginia, P.O. Box 800392

Charlottesville, VA 22908-0392 Telephone: (434) 924-5999 Email: <u>irbsbshelp@virginia.edu</u> Website: www.virginia.edu/vpr/irb/sbs

Website for Research Participants: <a href="http://www.virginia.edu/vpr/participants/">http://www.virginia.edu/vpr/participants/</a>

# **Electronic Signature Agreement:**

I agree to provide an electronic signature to document my consent.

| Teacher Printed Name: | |
|---|---|
| Signature: | Date: |
| I agree to partic | Study Agreement: ipate in the research study described above. |
| Teacher Printed Name: | |
| Signature: | Date: |
| School: | |
| Grade-Level Taught: | |

You will receive a copy of this form for your records.